CLINICAL TRIAL: NCT06823752
Title: A Dual Orexin Receptor Antagonist to Reduce Biomarkers of Neurodegeneration in Adults With Insomnia Disorder: a Randomised Placebo-controlled Cross-over Study.
Brief Title: A Dual Orexin Receptor Antagonist to Reduce Biomarkers of Neurodegeneration in Adults With Insomnia.
Acronym: Neuro-DORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Camilla Hoyos, Research Leader, Woolcock Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 16837
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Insomnia
Keywords: DORA; Tau; Beta Amyloid; Dementia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pick Disease of the Brain; Plaque, Amyloid; Dementia | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study staff (except the unblinded investigator) and the participants will be blinded. Blinding will be maintained by the use of identical containers and labels except for the patient identification code. The order of treatment will be secured in a password-protected data management system and known by the unblinded trial epidemiologist and a second designated person independent of the study team as back-up in the event of emergency unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dual Orexin Receptor Antagonist (DORA) (Experimental): 10mg Lemborexant tablet taken orally, nightly for two weeks
  Interventions: Drug: Lemborexant 10 MG
- Placebo (Placebo Comparator): Matching placebo tablet taken orally, nightly for two weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant 10 MG — An orally ingested tablet containing 10mg Lemborexant taken before bedtime. The investigational product is manufactured under Good Manufacturing Practice and is compliant with the TGA Therapeutic Order #101 that stipulates quality control requirements for capsule and pill-based products used in Australia.
  Other Names: Dayvigo
  Arms: Dual Orexin Receptor Antagonist (DORA)
Drug: Placebo — Placebo tablets will contain similar excipients without the active ingredient (Lemborexant) and manufactured under the same condition as the active. Placebo tablets, packs and instructions will be identical in every respect to enable the double-blind study design.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to explore the potential neuroprotective benefits of a dual orexin receptor antagonist (DORA) in adults with insomnia. The main questions it aims to answer are:

* Does the DORA reduce blood-based phosphorylated TAU181, in adults with insomnia, when compared to placebo
* Does the DORA reduce other blood-based biomarkers of neurodegeneration, including phosphorylated TAU217, amyloid beta 40:42 ratio, Neurofilament Light Chain (NFL) and Glial Fibrillary Acidic Protein (GFAP), when compared to placebo.

Participants will:

* Take 10mg Lemborexant nightly for two weeks
* Take a matching placebo nightly for two weeks
* Visit the research institute for a screening visit and for an overnight visit at the conclusion of each study drug treatment (3 visits in total).

DETAILED DESCRIPTION:
This is a randomised placebo-controlled cross-over study of a dual orexin receptor antagonist (DORA) versus placebo in adults with insomnia.

To be enrolled in the study, participants are required to complete an online pre-screening survey. Eligible participants will be directed to a separate webpage where they will be invited to review and download the Participant Information Sheet (PIS) and asked to provide their contact details and consent for a follow up call/email from the research team to book in a screening visit. At the screening visit the study team will explain the study to each participant and ensure they have had ample time prior to the visit to read and understand the PIS and have had the opportunity to ask any questions. The consent form will be signed by both the participant and a medical officer and participants will be randomised into their first treatment period; DORA (Lemborexant) or placebo.

Participants will take the treatment orally, nightly for 2 weeks. There will be a 2-4 week washout period between treatments. At the conclusion of both two-week treatment phases, participants will attend the laboratory for an overnight visit. The visit will take approximately 18 hours (including sleep time). During this visit, participants will partake in a number of assessments including HD-EEG, fNIRS, questionnaires and pupillometry. Participants will also have blood samples collected in the morning of the overnight study (hourly for four hours).

The study will recruit primarily through social media advertisements. The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Macquarie University, NSW, 2113, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia disorder as defined by the DSM-5 (difficulty initiating or maintaining sleep or waking up too early for at least 3 nights per week, for at least 3 months, with adequate opportunity and circumstances for sleep and at least one daytime impairment related to the sleep difficulty) and a score ≥15 on the ISI.
* Able to provide informed electronic consent.
* Fluent English literacy.
* Adults aged between 40-65 years.

Exclusion Criteria:

* People highly dependent on medical care as determined by a medical officer.
* Untreated moderate-severe sleep apnoea as diagnosed using in-home wrist oximetry (oxygen desaturation index>15, ongoing effectively treated sleep apnoea with insomnia will be allowed).
* Circadian disorders, narcolepsy, severe restless legs syndrome, and REM sleep behaviour disorder or uncontrolled psychiatric disorders.
* History of attempted suicide or current suicide ideation (indicated by a score >0 on Q9 of the Patient Health Questionnaire-9) at pre-screening.
* Objective cognitive decline measured by scoring ≤26 on the Montreal Cognitive Assessment (MoCA)
* Regular shift work, jet lag or trans-meridian travel (over 2h time difference) in the past week before randomisation.
* Pregnancy or lactation. Women will be advised to use contraception for the duration of the study and a urine pregnancy test will be performed when necessary.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical trial due to safety concerns or compliance with clinical study procedures.
* Currently participating in or has participated in a research study of an investigational agent or device within 4 weeks of enrolment.
* Concomitant use of medicines that are inhibitors (e.g., diltiazem, fluvoxamine, fluconazole, itraconazole, verapamil), or moderate to strong inducers of CYP3A4 (e.g., carbamazepine, modafinil, phenytoin, rifampicin, St John's Wort)
* Ongoing use of anti-psychotic medication, bosentan, efavirenz, etravirine, modafinil, rifampin, carbamazepine or illicit stimulants.
* Regular use of hypnotics (including melatonin, valerian, kava, benzodiazepines and Z-drugs), and other medications that can cause additive sedation (e.g. sedating antihistamines, tricyclic antidepressants, antipsychotics) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Regular use of psychostimulants (e.g., dexamfetamine, lisdexamfetamine, methylphenidate) or non-amphetamine psychostimulants (e.g., armodafinil, modafinil, atomoxetine) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Use of antidepressant medications for treatment of low mood for less than one year or dose changes (escalation or tapering) or change in antidepressant medications within the past year.
* Regular use opioids within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Ongoing use of THC- or CBD-containing products within 14 days prior to the start of the trial.
* Dependence or any other drug or alcohol dependence within the past two years (alcohol to be limited to no more than 2 standard drinks per day during trial period).
* Allergy to lactose.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Blood levels of TAU181 | 5 samples hourly for 4 hours after awakening in the morning of the overnight treatment period visits (approximately 7am-11am). We will test whether there is a difference between treatments over the time period.
  Morning blood-based phosphorylated TAU (standardised pTAU181:TAU181 ratio)

SECONDARY OUTCOMES:
Blood levels of TAU217 | 5 samples hourly for 4 hours after awakening in the morning of the overnight treatment period visits (approximately 7am-11am). We will test whether there is a difference between treatments over the time period.
  Morning blood-based phosphorylated TAU217, analysed within each participant.
Blood levels of Beta amyloid | 5 samples hourly for 4 hours after awakening in the morning of the overnight treatment period visits (approximately 7am-11am). We will test whether there is a difference between treatments over the time period.
  Morning blood-based Beta Amyloid 40:42 ratio, analysed within each participant.
Blood levels of NFL | 5 samples hourly for 4 hours after awakening in the morning of the overnight treatment period visits (approximately 7am-11am). We will test whether there is a difference between treatments over the time period.
  Morning blood-based Neurofilament Light Chain (NFL), analysed within each participant.
Blood levels of GFAP | 5 samples hourly for 4 hours after awakening in the morning of the overnight treatment period visits (approximately 7am-11am). We will test whether there is a difference between treatments over the time period.
  Morning blood-based Fibrillary Acidic Protein (GFAP), analysed within each participant.

OTHER OUTCOMES:
Absolute Electroencephalographic (EEG) Power During Non-Rapid Eye Movement (NREM) (stages 2 and 3) and REM sleep. | 14th night after treatment starts.
  High-density EEG, spectral power for frequency ranges low-delta: 0.5-1 Hz; delta: 1-4.5 Hz; theta: 4.5-8Hz; alpha: 8-12Hz; sigma: 12-15 Hz; beta: 15-25 Hz; gamma: 25-40 Hz. Absolute Electroencephalographic (EEG) Power During Non-Rapid Eye Movement (NREM) and REM sleep (12 statistical comparisons). Unit of measurement is μV^2.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Hoyos, MPH, PhD, Principal Investigator — Woolcock Institute of Medical Research; Brendon Yee, MBChB, FRACP, FCCP, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon reasonable request to the Principal Investigators.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Non-identifiable IPD will become available one year after the Actual Study Completion Date and will be available for ten years.
Access Criteria: A copy of the non-identifiable dataset may be requested by academic collaborators not affiliated with the WIMR through a data request form which outlines the investigators, aims and hypotheses, data to be included, a statistical analysis plan, ethics approval, and security measures. Contact the Coordinating Principal Investigator for access to data.